CLINICAL TRIAL: NCT05026385
Title: Targeted Knee Osteoarthritis Care for Adults With a BMI ≥35 kg/m2: the Prevention Of MusclE Loss in Osteoarthritis (P.O.M.E.L.O.) Feasibility and Pilot Randomized Trial
Brief Title: The POMELO (Prevention Of MusclE Loss in Osteoarthritis) Trial
Acronym: POMELO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: The Arthritis Society, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00107201
Record Dates: First submitted 2021-08-04; First posted 2021-08-30 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee; Obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive initial nutrition and exercise consultations with a Registered Dietitian (RD) and Clinical Exercise Physiologist (CEP) to personalize the study protocol and recommendations to their needs. The intervention period (3 months) includes: a) whole-body resistance training exercise sessions completed three-times per week (at-home with loaned equipment and/or in-person at the research gym); b) biweekly nutrition education provided through video conferencing; and c) biweekly OA self-management support provided through video conferencing.
  After the 3 month intervention, participants will receive bimonthly phone calls from a study staff member to encourage continued behavior changes during the 6 month maintenance phase.
  Interventions: Behavioral: Intervention
- Usual Care (No Intervention): The control group will follow standard care procedures, which includes their usual activities. The control group will receive bimonthly contact during the study period through phone calls with a study staff member to encourage retention. However no recommendations or advice on nutrition, exercise or self-management will be provided.

INTERVENTIONS:
Behavioral: Intervention — Targeted nutrition advice, progressive resistance training exercise, and self-management support
  Arms: Intervention

SUMMARY:
Treatment options for individuals who have advanced knee osteoarthritis (OA) and a body mass index (BMI) ≥35 kg/m2 are limited, and this patient population may be neglected in current clinical care pathways for OA management. These individuals are considered to be at high risk for complications with total knee arthroplasty (TKA), and as a result may not be eligible for this procedure unless they lose significant weight. However, there is limited evidence for endorsing weight loss as beneficial prior to TKA. Further, unsupervised weight loss could put patients at risk for muscle loss and development of sarcopenic obesity, a health condition that negatively impacts mobility and mortality. This suggests that weight loss might not be the primary treatment goal for this patient population. Integrated non-surgical treatment approaches are needed that can target the specific needs of this knee OA patient group. This study will examine the feasibility and acceptability of a personalized, multicomponent intervention, and its effects on body composition and physical function compared to usual care.

DETAILED DESCRIPTION:
The primary objectives of the POMELO study are to determine if a multicomponent behavioural intervention that includes personalized nutrition recommendations, progressive resistance training exercise, and chronic disease self-management support is feasible and acceptable for individuals living with advanced knee OA and a BMI ≥35 kg/m2. The secondary objectives are to assess potential effects of the intervention on muscle mass and physical function compared to usual care. The intervention is delivered over three months, followed by six months of ongoing maintenance support. Assessments are completed at baseline, interim (after the 3 month intervention phase), and at study end (after the 6 month maintenance phase) [for a total study period of 10 months]. This project will inform and influence the future development and implementation of more personalized knee OA treatment approaches for adults with a BMI ≥35 kg/m2 and reduce health disparities in access to effective care. Findings will also contribute to improved health outcomes for this vulnerable patient population, and enhanced delivery of health services by offering an alternative treatment pathway targeted to patient needs.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≥35 kg/m2
* unilateral or bilateral knee osteoarthritis (KL grade ≥2 and clinical symptoms)
* able to provide written, informed consent in English
* able to attend assessment appointments in Edmonton, Alberta
* have reliable and unlimited access to internet and a laptop, computer or tablet at home for access to videoconferencing sessions
* have space at home to complete exercises with equipment provided, or able to attend in-person exercise sessions

Exclusion Criteria:

* any medical conditions where participation in resistance exercise or nutrition adjustments are contraindicated
* neurological disorders (i.e. multiple sclerosis)
* post-traumatic OA with a fracture that impacts joint (secondary to injury or accident)
* rheumatoid arthritis
* prior bariatric surgery
* prior knee or hip replacement surgery
* recently (within 3 months) taken anabolic steroids or other muscle building compounds

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Per-protocol adherence (feasibility) | at interim (3 months)
  per-protocol adherence to the intervention >= 60%
Adverse events | at interim (3 months)
  rates of adverse events in the intervention and control arms
Study completion rates (feasibility) | at study completion (10 months)
  study completion rates >= 80%
Acceptability of Intervention Measure (AIM) score | at interim (3 months) and study completion (10 months)
  AIM scores compared between the intervention and control groups
Qualitative data on participants perceptions of acceptability | at interim (3 months) and study completion (10 months)
  qualitative data from open-ended survey and interview questions under each domain of the Theoretical Framework of Acceptability

SECONDARY OUTCOMES:
muscle mass | change from baseline to interim (3 months) and study completion (10 months)
  appendicular lean mass assessed by DXA
physical function (chair stands) | change from baseline to interim (3 months) and study completion (10 months)
  number of chair stands in 30 seconds
physical function (6MWT distance) | change from baseline to interim (3 months) and study completion (10 months)
  6MWT distance

OTHER OUTCOMES:
muscle quality | change from baseline to interim (3 months) and study completion (10 months)
  change in ultrasound-measured thigh muscle volume and echogenicity
fat mass | change from baseline to interim (3 months) and study completion (10 months)
  change in fat mass assessed by DXA
patient-reported health-related quality of life | change from baseline to interim (3 months) and study completion (10 months)
  change in quality of life assessed by EQ-5D
patient-reported arthritis-related pain and function | change from baseline to interim (3 months) and study completion (10 months)
  change in arthritis-related pain and function assessed by WOMAC
self-efficacy for managing chronic disease | change from baseline to interim (3 months) and study completion (10 months)
  change in self-efficacy scores assessed by PROMIS
lipid panel | change from baseline to interim (3 months) and study completion (10 months)
  change in blood assessed lipid panel (i.e. total cholesterol, LDL, HDL and triglycerides)
c-reactive protein | change from baseline to interim (3 months) and study completion (10 months)
  change in blood assessed c-reactive protein
insulin | change from baseline to interim (3 months) and study completion (10 months)
  change in blood assessed insulin
albumin | change from baseline to interim (3 months) and study completion (10 months)
  change in blood assessed albumin
liver enzymes | change from baseline to interim (3 months) and study completion (10 months)
  change in blood assessed liver enzymes (ALT and GGT)
glucose | change from baseline to interim (3 months) and study completion (10 months)
  change in blood assessed glucose
thyroid stimulating hormone | change from baseline to interim (3 months) and study completion (10 months)
  change in blood assessed thyroid stimulating hormone
resting energy expenditure | change from baseline to interim (3 months) and study completion (10 months)
  change in resting energy expenditure using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta; Mary Forhan, PhD, Principal Investigator — University of Toronto; Kristine Godziuk, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No